CLINICAL TRIAL: NCT02000960
Title: A Controlled N-of-1 Before-and-after Study to Determine Safety and Efficacy Triheptanoin in Patients With Glucose Transporter 1 Deficiency Syndrome
Brief Title: Pilot Study of Triheptanoin in Patients With Glucose Transporter 1 Deficiency Syndrome
Acronym: Glut1C7
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of British Columbia (Other)
Collaborators: Ultragenyx Pharmaceutical Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H13-03330; VGTPH001 (Other: Ultragenyx Pharmaceutical Inc.)
Record Dates: First submitted 2013-11-27; First posted 2013-12-04 (Estimated); Last update posted 2016-06-01 (Estimated); Status verified 2016-05

CONDITIONS: Glucose Transporter Type 1 Deficiency Syndrome
Keywords: Glut1 DS
MeSH Terms: conditions — Glut1 Deficiency Syndrome | interventions — triheptanoin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Triheptanoin (Experimental): All subjects will receive the study treatment which includes adding triheptanoin to the ketogenic diet with a goal intake of 35% total calories provided by triheptanoin (max 100 ml oil/day.
  Interventions: Drug: Triheptanoin

INTERVENTIONS:
Drug: Triheptanoin — Triheptanoin (C7 oil) is a triglyceride of the anaplerotic odd-chain fatty acid heptonate.
  Other Names: C7 oil

SUMMARY:
Glucose transporter deficiency syndrome (Glut1-DS) is a form of pediatric epilepsy caused by a genetic mutation that disrupts the body's ability to process food from the child's diet into sugar (energy) needed to support brain function. Children with Glut1-DS experience seizures that are not controlled by anticonvulsant medications, as well as delays in cognitive and motor development. Currently, Glut1-DS is treated with the ketogenic diet, a high-fat, low-sugar diet that provides the brain with an alternate source of energy. Despite the significant improvement of seizures upon this diet, seizure control is incomplete in a majority of children, and they continue to experience problems with brain development. Our team of researchers and clinicians with expertise in metabolic diseases, neurology, pediatrics, biochemistry, and genetics believes that there is an opportunity to achieve CURE's goal of "No Seizures/No Side Effects" for children with Glut1-DS by investigating the use of a new treatment option that is designed to compensate for the underlying biochemical deficiency thought to contribute both to the seizures and to the impaired brain development associated with Glut1-DS. The proposed treatment involves incorporating a special type of oil, called triheptanoin, into the ketogenic diet as a way to make up for a specific biochemical deficit affecting kids with Glut1-DS that the standard ketogenic diet fails to address. Our goal is to do a pilot study to test the safety and effectiveness of this promising new treatment option in a small group of children with Glut1-DS.

DETAILED DESCRIPTION:
BACKGROUND: Glucose transporter type 1 deficiency syndrome (Glut1-DS) is a metabolic epileptic encephalopathy caused by defects in the cerebral glucose transporter GLUT1. It is characterized by infantile seizures refractory to anticonvulsants, deceleration of head growth, and delays in mental and motor development. Low brain glucose and subsequent energy deficiency is considered the major pathogenic factor causing seizures. The ketogenic diet (KD) is the only causal treatment available for Glut1-DS, and its therapeutic effect resides in its ability to provide an alternate source of energy for the brain. However, seizure control with KD is not complete in many patients and the long-term cognitive outcome is not optimal. Biochemically, these observations can be explained by a lack of energy for metabolic functions provided by pathways derived exclusively from glucose, which the alternate energy from the KD fails to supplement.

HYPOTHESIS: We hypothesize that an anaplerotic agent adjunct to KD may be effective for controlling seizures and improving cognitive outcomes in children with Glut1-DS. Triheptanoin (C7) is a triglyceride containing the odd chain C7 (heptanoic) fatty acid, which occurs only in limited amounts in the natural diet. It improves the oxidation of acetyl CoA by the tricarbonic acid (TCA) cycle, leading to subsequent oxidative phosporylation by the electron transport chain to produce sufficient ATP for energy utilization. It also provides the TCA intermediates alpha ketoglutarate and oxaloacetate, which are important precursors for the neurotransmitters glutamate, GABA, and aspartate. Therefore, we expect these metabolic effects will enhance seizure control and/or neurodevelopmental function.

SPECIFIC AIMS: We aim to generate preliminary evidence on 1) the safety, 2) the clinical, and 3) the biochemical effects of C7 as an add on therapy in GLUT1-DS patients with inadequate response to ketogenic diet.

RESEARCH PLAN: To generate preliminary data and a better understanding of the precise biochemical mechanism of this novel treatment, we will conduct a pilot/proof of concept study using an open-label n-of-1 trial with 'an interrupted time-series before and after' design. We plan to enrol 3 Glut1-DS patients with incomplete seizure control, and the n-of-1 study design will help provide a distinct effectiveness estimate of C7 in each individual patient. As each participant acts as his/her own control, this design also supports an evidence-based, personalized medicine approach to treatment.

SIGNIFICANCE: If successful, this personalized treatment approach may be extended to GLUT1-DS patients with other symptoms refractory to the KD, or those who cannot tolerate the diet, and ultimately will serve as a model for eliminating seizures and side effects in other medically refractory epilepsies. The data generated with this study will be essential to design future trials for a larger number of Glut1-DS patients to create high-grade evidence.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of Glut1-DS with mutation(s) in SLC2A1 gene.
* Male or female age 1-18 years.
* Glut1-DS is currently managed with ketogenic diet for a minimum of 4 months prior to baseline visit and patient is willing to maintain this diet for the study duration..
* Inadequate response to ketogenic diet defined by clinical 'breakthrough seizures', confirmed by EEG and at least 1 clinical seizure episode documented in the seizure logbook during the baseline period.
* For participants taking anticonvulsants for their seizures, anti-seizure medication should not be changed at least 4 weeks prior to starting triheptanoin treatment and the participant is willing to maintain the same dosing of all medication(s) during study participation.
* Willing and able to provide written informed consent by parent(s) or guardian(s) or assent by the participant, depending on the age, after the nature of the study has been explained, and prior to any research related-procedures.

Exclusion Criteria:

* Participants with medium chain acyl-CoA dehydrogenase (MCAD) and propionyl CoA carboxylase (PCC) deficiency will be excluded from the study as MCAD and PCC are required for triheptanoin metabolism.
* A known allergy or sensitivity to any component of triheptanoin.
* The participant is using valproate for controlling his/her seizures. They are eligible for the study, if they had not taken valproate within 3 weeks prior to baseline visit and willing to not take it for the entire study duration. Valproate is an AED that partially inhibits the TCA cycle via alpha-ketoglutarate dehydrogenase, and should not be administered to subjects taking triheptanoin.
* Participant has any condition or situation which, in the investigator's opinion, places the patient at significant risk of adverse events, or may interfere significantly with their participation and compliance in the study.

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 3 (Estimated)
Dates: Start 2014-04; Primary Completion 2016-02 (Actual); Study Completion 2016-10 (Estimated)

PRIMARY OUTCOMES:
Seizure Control | 8 months
  Complete seizure control (measured using seizure log book completed by the parents; defined by absence of clinical seizures and normalization of the EEG)

SECONDARY OUTCOMES:
Biochemical markers | 8 months
  Specific biochemical markers and metabolomics analysis to determine the metabolic fate of the administered Triheptanoate will be done at Case Western Reserve University, Cleveland.
  Markers:
  Urine:
  TCA compounds: Succinate, fumarate, alphaketoglutarate Anaplerotic precursors: Propionate Ketone bodies: Betahydroxybutyrate, acetoacetate
  Blood:
  Aminoacids: Glutamate, gluatamine, alanine Acylcarnitine/propionylcarnitine Beta hydroxypentanoate, beta ketopentanoate;
  CSF:
  Aminoacids: Glutamate, gluatamine, alanine
Neurodevelopmental function | 8 months
  This will be measured by a psychologist using age-appropriate measurement scales from the NIH Toolbox (http://www.nihtoolbox.org).
Movement Disorder | 8 months
  assessed by neurological exam, Movement Disorder Childhood Rating Scale1 and tests from NIH Toolbox

OTHER OUTCOMES:
Seizure Frequency | 8 months
  Median percent reduction in frequency of seizures from baseline from seizure log book.
Clinical Global Impression-Improvement Scale | 8 months
  Treatment response measured by Clinical Global Impression-Improvement Scale
Patient specific outcomes of interest | 8 months
  Patient specific outcomes of interest measured by Goal Attainment Scale

CONTACTS AND LOCATIONS:
Overall Officials: Sylvia Stockler, Principal Investigator — The University of British Columbia/BC Children's Hospital
Locations (1):
- BC Children's Hospital, Vancouver, British Columbia, Canada